CLINICAL TRIAL: NCT05683847
Title: Effects of EpilepsiNett - User Controlled Follow-up Developed by a Nationwide, Multidisciplinary Network of Epilepsy Experts
Brief Title: User Controlled Follow-up of Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Haukeland University Hospital (Other); Oslo University Hospital (Other); University of Oslo (Other); University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: REK 30892
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy
Keywords: epilepsy; patient reported outcome measures; PROM; outpatient follow-up
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with epilepsy: User controlled epilepsy follow-up by means of digital patient reported outcome measures (PROM).
  Interventions: Other: User controlled epilepsy follow-up by means of patient reported outcome measures (PROM)

INTERVENTIONS:
Other: User controlled epilepsy follow-up by means of patient reported outcome measures (PROM) — Whenever they want to, but minimum every six months, users respond to standardized follow-up questions developed by the experts of EpilepsiNett. This ensures that a broader range of topics are covered, not just those related to seizures and adverse events. The incoming responses are handled by a trained epilepsy nurse, who contact the patient when needed, consulting the responsible medical doctor when needed. If current issues cannot be solved by telephonic contact with the epilepsy nurse and/or responsible medical doctor, the patient is offered an appointment at the outpatient clinic.

SUMMARY:
In December 2019 Vestre Viken Hospital Trust implemented user controlled epilepsy follow-up. Patients receive follow-up questions digitally twice yearly. The questionnaire was made by a multidisciplinary national network of epilepsy experts (EpilepsiNett). Responses to the questionnaire are controlled by an epilepsy nurse, and further follow-up is based on this. Data collected for user controlled follow-up will be matched with data from national registries, investigating whether this type of follow-up influences the patients' clinical course and/or the hospital's and society's use of resources.

DETAILED DESCRIPTION:
Vestre Viken Hospital Trust implemented user controlled follow-up by means of PROMs reported digitally in December 2019. Whenever they want to, but minimum every six months, users respond to standardized follow-up questions developed by the experts of EpilepsiNett, a multidisciplinary national network of epilepsy researchers. This ensures that a broader range of topics are covered, not just those related to seizures and adverse events. The incoming responses are handled by a trained epilepsy nurse, who contact the patient when needed, consulting the responsible medical doctor when needed. If current issues cannot be solved by telephonic contact with the epilepsy nurse and/or responsible medical doctor, the patient is offered an appointment at the outpatient clinic.

In collaboration with the Norwegian Institute of Public Health (FHI), the aim is to make user controlled epilepsy follow-up by means of PROMs a national standard for epilepsy care in Norway. In order to achieve this, data and documentation of its effects is crucial.

From Vestre Viken's internal reporting system, the investigators will extract the number of consultations in the outpatient clinic of neurology with a diagnostic code of epilepsy (ICD-10 G40.0-G40.9) for the years 2017-2019 and calculate a yearly average (total and per patient) of epilepsy-related visits before implementation of user-controlled epilepsy follow-up (Dec. 2019). The investigators will then extract the same data for the years 2020, 2021 and 2022 and compare to the mentioned average. Prevalence and incidence of epilepsy are expected to be stable across these years, but visits in the outpatient clinic are expected to be lower in the pandemic years of 2020 and 2021. Thus, the results from 2022 will be important. The same calculations will be done for visits to the emergency room outpatient clinic, and for emergency hospital admissions.

Data will be extracted from the digitally registered PROMs at Drammen Hospital (Dec. 2019-Dec. 2022) and Haukeland University Hospital (Dec. 2020-Dec. 2022). The investigators will analyze adherence, seizure frequency and quality of life in all patients included in user controlled epilepsy follow-up at baseline, and after two years of such follow-up.

Data from national registries will also be used. EpilepsiNett has received a large registry based data package, combining variables several Norwegian health registries. The connection of data from the different registries will be done by The Norwegian Prescription Database, including a file with IDs of the patients included in user controlled epilepsy follow-up, and delivers a pseudonymized file to the head of research of EpilepsiNett, who controls and distributes the data to our researchers.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of epilepsy. Age>18 years.

Exclusion Criteria:

Not able to handle the digital tools required for this type of follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults with a diagnosis of epilepsy visiting the outpatient clinic or the Dep. of Neurology in Vestre Viken Hospital Trust.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of visits to the outpatient clinic before and after implementation of user controlled epilepsy follow-up | 2 years
  We hypothesize a decline in outpatient clinic visits for the people enrolled in user controlled epilepsy follow-up
Number of emergency hospitalizations before and after implementation of user controlled epilepsy follow-up | 2 years
  We hypothesize a decline in emergency hospitalization for the people enrolled in user controlled epilepsy follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marte Syvertsen, PhD, Study Chair — Vestre Viken Hospital Trust
Locations (1):
- Drammen Hospital, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No